CLINICAL TRIAL: NCT04814017
Title: Effectiveness of Radial Shock-wave Therapy Combined With Self-stretching Exercises in Patients With Myofascial Pain Syndrome
Brief Title: Effectiveness of Shock-wave Therapy in Patients With Myofascial Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Fatma Uguz Selcuk, Principal Investigator, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24.01.2013/2
Record Dates: First submitted 2021-03-14; First posted 2021-03-24 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Myofascial Pain Syndrome; Chronic Pain
Keywords: Physiotherapy; shock wave therapy; stretching exercises
MeSH Terms: conditions — Myofascial Pain Syndromes; Chronic Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radial shock-wave group (Experimental): Group I (15 subjects) received radial shock-wave application one times a week for six weeks and home based stretching exercises.
  Interventions: Procedure: Radial Shock-Wave Therapy
- Control (Experimental): Group II (15 subjects) received home based stretching exercises for six weeks.
  Interventions: Procedure: Control

INTERVENTIONS:
Procedure: Radial Shock-Wave Therapy — Radial shock-wave therapy was applied in 1.0-4.0 bar intensity, 10-15 hz frequency interval. 300-700 pulse for a trigger point, 1500-3000 pulse for a muscle. Intensity, frequency and pulse increased every session regularly beginning from minimal taking patients tolerance into consideration. Trigger points in the upper, middle and lower trapezius, supraspinatus, infraspinatus and levator scapula muscles were treated. Neck and upper back muscle static stretching exercises were teached to patients as home exercise program. The patients were asked to do each stretching exercise given as a home-based program every day, 3 times a day and 3 repetitions. The exercise program consisted of static neck lateral flexors stretching, shoulder posterior capsule stretching and apley stretching exercises. Exercise booklets were prepared and given to the patients.
  Arms: Radial shock-wave group
Procedure: Control — Neck and upper back muscle static stretching exercises were teached to patients as home exercise program. The patients were asked to do each stretching exercise given as a home-based program every day, 3 times a day and 3 repetitions. The exercise program consisted of static neck lateral flexors stretching, shoulder posterior capsule stretching and apley stretching exercises. Exercise booklets were prepared and given to the patients.
  Arms: Control

SUMMARY:
30 patients with chronic cervical myofascial pain (4 males, 26 females) aged between 25 to 57 years (with average age 41,20±10,23 years) were included the study.

Participants were divided into two groups as intervention group (n=15) and control group (n=15). Patients in intervention group received radial shock-wave application one times a week for six weeks and home based stretching exercises. Patients in control group (CG) received home based stretching exercises. Rest and activity pain (Visual Analog Scale), pressure pain threshold (PPT), cervical range of motion (CROM) and disability (Neck Disability Index) were assessed at baseline and after the treatment.

DETAILED DESCRIPTION:
Thirty-four cervical MPS patients aged between 25-57 years (average age: 41,20±10,23 years) who diagnosed cervical MPS (myofascial pain syndrome), had cervical MPS for 6 months and who had at least one trigger point on their cervical, back and shoulder muscles were included to this study.

Thirty-four participant were included to the study. Taking into consideration including and excluding factors 34 participants divided into two groups: intervention shock-wave therapy group, control group. Because of several private reason (not attending treatment regularly and not participating in the final evaluations), 4 participant were excluded from study.

All assessments done by the same physiotherapist (FU) before the first session and one week after the last treatment session. Demographic data of participants recorded by using a form at the baseline of the study.

Patients in the intervention group (n=15) received 6 sessions radial shock wave treatment once a week during 6 weeks. During the treatment, the patients sat on chairs and supported their upper bodies with a pillow on the bed. Ultrasound gel was applied to the application area. Radial shock-wave therapy was applied to each trigger point in the preliminary evaluation. The muscles related trigger points were stretched position during the application. Radial shock-wave therapy was applied in 1.0-4.0 bar intensity, 10-15 hz frequency interval. 300-700 pulse for a trigger point, 1500-3000 pulse for a muscle. Intensity, frequency and pulse increased every session regularly beginning from minimal taking patients tolerance into consideration. Trigger points in the upper, middle and lower trapezius, supraspinatus, infraspinatus and levator scapulae muscles were treated.

Neck and upper back muscle static stretching exercises were teached to patients in the both groups as home exercise program. The patients were asked to do each stretching exercise given as a home-based program every day, 3 times a day and 3 repetitions. The exercise program consisted of static neck lateral flexors stretching, shoulder posterior capsule stretching and apley stretching exercises. Exercise booklets were prepared and given to the patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed cervical MPS
* Have cervical MPS for at least 6 months.
* Patients who has at least one trigger points on their cervical, back and shoulder muscles.

Exclusion Criteria:

* Fibromyalgia diagnosed patients in reference to 1990 ACR criteria.
* Patients who has characteristic cervical disc degeneration, radiculopathy, myelopathy.
* Patients who has cervical fracture, tumor, infection, malign, psychiatric and systemic illness.
* Patients who had an operation because of cervical problem.
* Patients who is treated with another treatment technique at the same time.
* Being pregnant

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-01-28 (Actual); Primary Completion 2013-04-10 (Actual); Study Completion 2013-06-30 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | Baseline
  Pain intensity was measured using a Visual Analogue Scale (VAS) measuring 10 cm (0: I have no pain, 10: I have an intolerable pain).
Cervical Range of Motion | Baseline
  Cervical range of motion (CROM) tool was used to assess cervical range of motion. Measurements were repeated three times in flexion, extension, rotation and lateral flexion directions.
Disability | Baseline
  Turkish version of Neck Disability Index (NDI) was used to assess the disability caused by neck pain.
Pressure pain threshold (PPT) | Baseline
  Digital pressure algometer applied to patients active trigger points.

SECONDARY OUTCOMES:
Pain Intensity | 6 weeks
  Pain intensity was measured using a Visual Analogue Scale (VAS) measuring 10 cm (0: I have no pain, 10: I have an intolerable pain).
Cervical Range of Motion | 6 weeks
  Cervical range of motion (CROM) tool was used to assess cervical range of motion. Measurements were repeated three times in flexion, extension, rotation and lateral flexion directions.
Disability | 6 weeks
  Turkish version of Neck Disability Index (NDI) was used to assess the disability caused by neck pain.
Pressure pain threshold (PPT) | 6 weeks
  Digital pressure algometer applied to patients active trigger points.

CONTACTS AND LOCATIONS:
Overall Officials: Aysenur OYMAK SOYSAL, Dr., Study Chair — Saraykoy Vocational School; Erol Ozen, Dr., Study Chair — Denizli Private Health Hospital
Locations (1):
- Silivri Public Hospital, Istanbul, Silivri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Because there is no web site to share my data

REFERENCES:
- [Result] Kiraly M, Bender T, Hodosi K. Comparative study of shockwave therapy and low-level laser therapy effects in patients with myofascial pain syndrome of the trapezius. Rheumatol Int. 2018 Nov;38(11):2045-2052. doi: 10.1007/s00296-018-4134-x. Epub 2018 Aug 31. PMID 30171341
- [Result] Williams MA, Williamson E, Gates S, Cooke MW. Reproducibility of the cervical range of motion (CROM) device for individuals with sub-acute whiplash associated disorders. Eur Spine J. 2012 May;21(5):872-8. doi: 10.1007/s00586-011-2096-8. Epub 2011 Dec 3. PMID 22139052
- [Result] Aslan E, Karaduman A, Yakut Y, Aras B, Simsek IE, Yagly N. The cultural adaptation, reliability and validity of neck disability index in patients with neck pain: a Turkish version study. Spine (Phila Pa 1976). 2008 May 15;33(11):E362-5. doi: 10.1097/BRS.0b013e31817144e1. PMID 18469684
- [Result] Ay S, Dogan SK, Evcik D, Baser OC. Comparison the efficacy of phonophoresis and ultrasound therapy in myofascial pain syndrome. Rheumatol Int. 2011 Sep;31(9):1203-8. doi: 10.1007/s00296-010-1419-0. Epub 2010 Mar 31. PMID 20354859